CLINICAL TRIAL: NCT04913025
Title: REduced Frequency ImmuNE Checkpoint Inhibition in Cancers: A Multi Arm Phase II Basket Protocol Testing Reduced Intensity Immunotherapy Across Different Cancers
Brief Title: REduced Frequency ImmuNE Checkpoint Inhibition in Cancers
Acronym: REFINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: JP Moulton Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RF01; 2021-002060-47 (EudraCT Number)
Record Dates: First submitted 2021-05-13; First posted 2021-06-04 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Renal Cell Carcinoma; Melanoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma | interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard interval (Active Comparator): Standard of care regimen Nivolumab administered as an approximate 60-minute IV infusion, as a flat dose of 480mg once every 4 weeks OR Pembrolizumab administered as an approximate 60-minute IV infusion, as a flat dose of 400mg once every 6 weeks
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab
- Extended interval (Experimental): Nivolumab administered as an approximate 60-minute IV infusion, as a flat dose of 480mg once every 8 weeks OR Pembrolizumab administered as an approximate 60-minute IV infusion, as a flat dose of 400mg once every 12 weeks
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nivolumab — 60-minute IV infusion, as a flat dose of 480mg
Drug: Pembrolizumab — 60-minute IV infusion, as a flat dose of 400mg

SUMMARY:
The REFINE trial aims to asses whether giving an immunotherapy drug less-often to patients with advanced cancer, results in fewer side effects whilst continuing to be an effective treatment. The question will be assessed in different tumour types by means of different cohorts within an overarching trial protocol.

DETAILED DESCRIPTION:
In stage I eligible participants will be randomly assigned to either the standard interval (either 4 or 6 weeks) or the extended interval (either 8 or 12 weeks) following an initial 12 weeks of standard of care immunotherapy. Disease recurrence and survival will be assessed, along with quality of life and health economic outcomes. The trial includes a feasibility outcome by which recruitment feasibility will be assessed.

Immunotherapy drugs are a standard treatment option for advanced kidney cancer, melanoma, and some lung cancers. These drugs work by stimulating the body's own immune system to fight against cancer cells. Clinical trials have proven the effectiveness of immunotherapy drugs, such as ipilimumab, nivolumab or pembrolizumab, in the treatment of different cancers. However the best way to give these drugs is not known.

ELIGIBILITY:
Common Inclusion Criteria:

* WHO Performance Status 0 or 1.
* Patients with locally advanced or metastatic cancer whose clinician has determined they are candidates for treatment with standard of care immune checkpoint inhibitor.- Patients aged ≥18years.
* Adequate normal organ and marrow function:

  1. Haemoglobin ≥9.0g/dL (transfusions will be allowed within 2 weeks prior to randomisation in order to achieve the entry criteria).
  2. Absolute neutrophil count (ANC) ≥1.5 x 109/L (≥1500 per mm3).
  3. Platelet count ≥100 x 109/L (≥100,000 per mm3).
  4. Bilirubin ≤1.5 x ULN (This will not apply to subjects with confirmed Gilbert's syndrome (i.e., persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), who will be considered eligible only in consultation with their physician).
  5. AST/ALT ≤3 x ULN.
  6. eGFR >40mL/min by CKD-EPI formula .
* Both men and women enrolled in this trial must be in agreement with trial policy on contraception during the treatment phase of the study. Egg donation, sperm donation and breastfeeding must be avoided.
* Evidence of post-menopausal status or negative serum HCG pregnancy test for female pre/peri-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  1. Women <50 years of age will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormone treatments and if they have luteinising hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilisation (bilateral oophorectomy or hysterectomy).
  2. Women ≥50 years of age will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilisation (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

Renal Cohort Inclusion Criteria:

* Patients with unresectable locally-advanced or metastatic renal cell carcinoma (including clear cell and papillary histologies).
* Intermediate or poor risk as defined in the International Metastatic Renal Cell Carcinoma Database Consortium criteria.
* Patient has received induction ipilimumab (all four doses) and nivolumab as first-line treatment as planned.
* Due to commence maintenance nivolumab with no evidence of progression (i.e. response or stable disease on cross sectional imaging on completion of initial 12 weeks treatment with ICI).

Melanoma Cohort Inclusion Criteria

* Patients with locally-advanced or metastatic melanoma.
* Patients have received single agent pembrolizumab first-line for 3 months, with no evidence of progression (i.e. response or stable disease) on cross sectional imaging 12 weeks after initiation of ICI, and due to commence maintenance pembrolizumab every 6 weeks.

or Patients have received induction ipilimumab 1mg/kg and nivolumab 3mg/kg as first-line treatment, and due to commence maintenance nivolumab with no evidence of progression (i.e. response or stable disease) on cross sectional imaging 12 weeks after initiation of ICI.

Exclusion Criteria:

* Patients who have received ICI in a prior line of treatment.
* Patients whose planned treatment is the combination of anti-PD-1 and tyrosine kinase inhibitor e.g. pembrolizumab+axitinib or the combination of traditional cytotoxic chemotherapy and anti-PD-1.
* Patients with unresolved/untreated immune-related adverse events arising during the first 3 months treatment with standard of care ICI.
* History of another previous malignancy, except for:

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP.
  2. Adequately treated non-melanoma skin cancer without evidence of disease.
  3. Adequately treated carcinoma in situ without evidence of disease.
  4. Superficial bladder cancer.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Current or prior use of immunosuppressive medication within 14 days of starting trial treatment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10mg/day of prednisone, or an equivalent corticosteroid.
* Active infection including:

  1. Tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).
  2. Hepatitis B (known positive HBV surface antigen (HBsAg) result). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
  3. Hepatitis C. Note: Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
  4. Human immunodeficiency virus (positive HIV 1/2 antibodies).
* Receipt of a live attenuated vaccine within 30 days prior to the start of treatment.

Note: Patients, if enrolled, should not receive a live vaccine while receiving immune checkpoint inhibitor and up to 30 days after the last dose of immune checkpoint inhibitor.

* Known allergy or hypersensitivity to immune checkpoint inhibitor.
* Pregnant or breastfeeding patients.
* Uncontrolled adrenal insufficiency.
* Any serious or uncontrolled medical or psychiatric disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, interfere with participation and/or compliance in the trial, or interfere with the interpretation of study results.
* Participants who have undergone any prior systemic anti-cancer treatment (previous participation in adjuvant studies allowed, providing the patient was on the observation/ placebo arm - this may require un-blinding of the patient).
* Untreated brain metastases or brain metastases treated only with whole brain radiotherapy. (Patients are eligible if previous brain metastases treated with complete surgical resection, Stereotactic Brain Radiation Therapy (SBRT), or gamma knife with no subsequent evidence of progression and asymptomatic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year 9 months follow-up
  Time to event

SECONDARY OUTCOMES:
Overall survival | 1 year 9 months follow-up
  Measured from date of randomisation until date of death or last follow-up
Quality of Life (QoL) - Generic | 1 year 9 months follow-up
  EQ-5D-5L questionnaire to assess generic quality of life
Treatment-related toxicity | 1 year 9 months follow-up
  Measured using severity of all AEs and/or ARs (serious and non-serious) with the toxicity scales in NCI CTCAE v5.0 reviewed at the end of each stage and reported until trial closure
Mean incremental cost per patient | 1 year 9 months follow-up
  Measured using unit costs from NHS Reference Costs, Personal Social Services Research Unit (PSSRU) and British National Formulary (BNF) prices, and applying them to health and social care resource use collected via the Client Service Receipt Inventory (CSRI), intervention medication CRF, additional treatment logs, and concomitant medication CRF, every 12 weeks starting at baseline, calculating the cost and taking the difference between arms to calculate mean incremental cost per patient (bootstrapped regression, adjusting for baseline values, jointly with QALYs).
Mean incremental quality-adjusted life-years (QALYs) per patient | 1 year 9 months follow-up
  Measured using utility scores calculated from EQ-5D-5L questionnaire responses collected every 12 weeks starting at baseline, and applying them to the relevant period of follow-up to calculate quality-adjusted life-years (QALYs), and taking the difference between arms to calculate mean incremental QALYs per patient (bootstrapped regression, adjusting for baseline values, jointly with costs).
Cost-utility analysis | 1 year 9 months follow-up
  Assessing cost-effectiveness of reduced vs. standard frequency administration with summary result expressed as the incremental cost-effectiveness ratio (ICER), i.e. incremental cost per QALY gained, calculated by dividing incremental costs by incremental QALYs; with sensitivity analysis expressed via cost-effectiveness planes and cost-effectiveness acceptability curves to indicate probability that the intervention is cost-effective compared to the standard of care for a range of values of the cost-effectiveness threshold
Feasibility of recruitment to each cohort | 1 year 9 months follow-up
  Measured by sites completing screening logs to identify number of treatment cycles
Quality of Life (QoL) - Cancer-specific | 1 year 9 months follow-up
  EORTC QLQ-C30 questionnaire to assess cancer-specific quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Gilbert, Study Director — MRC CTU at UCL
Locations (3):
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Castle Hill Hospital, Hull
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merrick S, Nankivell M, Quartagno M, Clarke CS, Joharatnam-Hogan N, Waddell T, O'Carrigan B, Seckl M, Ghorani E, Banks E, Edmonds K, Bray G, Woodward R, Bennett R, Badrock J, Hudson W, Langley RE, Vasudev N, Pickering L, Gilbert DC. REFINE (REduced Frequency ImmuNE checkpoint inhibition in cancers): A multi-arm phase II basket trial testing reduced intensity immunotherapy across different cancers. Contemp Clin Trials. 2023 Jan;124:107030. doi: 10.1016/j.cct.2022.107030. Epub 2022 Nov 26. PMID 36519749